CLINICAL TRIAL: NCT04238468
Title: Scar Tissue Analysis After Intraoperative Intradermal Application of Stromal Vascular Fraction Cells Into Suture Line
Brief Title: Scar Tissue Analysis After Intraoperative Application of Stromal Vascular Fraction Cells Into Suture Line
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Katarina Zivec (Other)
Responsible Party: Sponsor-Investigator, Katarina Zivec, Principal Investigator, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSVF
Record Dates: First submitted 2020-01-18; First posted 2020-01-23 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Wound Heal; Scar; Hypertrophic Scar; Delayed Wound Healing
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient, investigator, outcome assessor will be blinded for which side of the scar was injected with stromal vascular fraction. Only the surgeon will know which site was injected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradermal injection of stromal vascular fraction (Experimental): Most lateral 5 cm of abdominal donor site will be injected with stromal vascular fraction just after the wound is closed.
  Interventions: Procedure: Intradermal stromal vascular fraction injection
- control (No Intervention): Most contralateral 5 cm of abdominal donor site will serve as control.

INTERVENTIONS:
Procedure: Intradermal stromal vascular fraction injection — After flank liposuction, lipoaspirate will be processed by enzymatic digestion, thus stromal vascular fraction will be isolated. Just after the wound is closed the stromal vascular fraction diluted in normal saline (5ml) will be injected intradermally on one site.
  Arms: Intradermal injection of stromal vascular fraction

SUMMARY:
The study will evaluate the effect of intradermal injection of stromal vascular fraction into suture line on wound healing and scarring.

DETAILED DESCRIPTION:
Patients undergoing primary or secondary Deep Inferior Epigastric Perforator (DIEP) flap breast reconstruction will be included in this monocentric, randomised, controlled, double-blinded study.

After bilateral flank liposuction, the fat will be processed by a special protocol with enzymatic digestion. Stromal vascular fraction will be isolated and injected intradermally just after wound closure into one site of surgical wound (most lateral 5 cm) at the DIEP flap donor site. The other site of DIEP flap donor site (most lateral 5 cm) will serve as a control. Part of stromal vascular fraction will be analysed by flow cytometry for the viability and cell specification. Ten months after DIEP flap surgery the scars at both sites (control and injected site) will be excised and analysed histologically. At that time photographs will be taken and scars will be analysed by Patient and Observer Assesment Scale (POSAS).

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients scheduled for primary or secondary DIEP flap breast reconstruction

Exclusion Criteria:

* BMI
* age
* immunosuppressive disease

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-10-10 (Estimated)

PRIMARY OUTCOMES:
Analysis of stromal vascular fraction by flow cytometry | 2 hours
  Cell viability and cell type specification of stromal vascular fraction will be evaluated by flow cytometry.
Histological analysis of epidermal thickness of scar tissue | 10 months
  Epidermal thickens of scar tissue on the injected and control site will be compared.
Histological analysis of rete ridges of scar tissue | 10 months
  Number of rete ridges of scar tissue on the injected and control site will be compared.
Histological quantification of elastin of scar tissue. | 10 months
  Quantification of elastin of scar tissue will be compared on the injected and control site.
Histological quantification of vascularity in scar tissue | 10 months
  Vascularity will be histologically quantified and compared on the injected and control site.
Histological quantification of inflammatory cells in scar tissue | 10 months
  Inflammatory cells will be histologically quantified and compared on the injected and control site.
Clinical outcome by the use of Patient and Observer Scar Assessment Scale (POSAS) | 10 months
  Scar will be evaluated by the Patient and Observer Scar Assessment Scale. The POSAS consists of two parts: a Patient Scale and an Observer Scale. Both scales contain six items that are scored numerically and make up a 'Total Score' of the Patient and Observer Scale. The sum altogether will give the 'Total Score' of the POSAS. Besides the 10-step scale, category boxes are available to score nominal parameters (e.g. type of colour). Moreover, the patient and observer also score their 'Overall Opinion'.

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Zivec, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia